CLINICAL TRIAL: NCT06910293
Title: Whole-Brain Dynamics in the Natural Menstrual Cycle vs. an Ovarian Stimulated Cycle: Impact of Hormonal Fluctuations on Healthy Women Undergoing Ovarian Stimulation
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: Khalifa University for Science and Technology (Other); New York University Abu Dhabi (Other)
Responsible Party: Principal Investigator, Dr. Raquel Del Gallego Bonilla, Head Clinical Data Management Unit, ART Fertility Clinics LLC
Other Study IDs: 22502-ABU-006-RDG
Record Dates: First submitted 2025-03-10; First posted 2025-04-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Neural Activity; Brain Function; Neurodynamics; Brain Connectivity
Keywords: Menstrual Cycle; Ovarian Stimulated Cycle; Endocrine Profile; neural activity; neurodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — The first visit will include an additional genetic testing, to perform association analysis between genetic and neuroimaging and fertility data. The investigator will collect saliva samples from the study participants during their visit to NYUAD using a standard saliva collection kit. Samples will be stored on the facility freezers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young (age range 25-35), healthy , who want to undergo ovarian stimulation for oocyte vitrification.: - Initial Assessment of Volunteers for Inclusion in the study.
  Once included, volunteers will need to be assessed 8 times during the study period, with 6 fMRI scans:
  * Natural menstrual cycle (depending on cycle duration: around 26-35 days)
    1. Basal (day 2-3 of the menstrual cycle)
    2. Monitoring of follicle growth (no fMRI at these monitoring dates)
    3. Day of LH surge +/-1 day (around day 14, 2-3 hormonal checks will be needed to identify Ovulation Day)
    4. Mid-Luteal (6-7 days after ovulation)
  * Stimulated Cycle 5. Basal (day 2-3 of the menstrual cycle) 6. Standard monitoring during ovarian stimulation (no fMRI at these monitoring dates) 7. Day between administration of final oocyte maturation & Oocyte Pick-Up (OPU) 8. Mid-luteal (6-7 days after OPU)
  Every stage will include a blood test for hormonal evaluation, vaginal ultrasound for follicular count & sizing, administration of MRI protocol. The first visit will include buccal swab.
  Interventions: Diagnostic Test: Functional Magnetic resonance imaging will be done on day 2 or 3 of the menstrual cycle, trigger-shot and egg retrieval.

INTERVENTIONS:
Diagnostic Test: Functional Magnetic resonance imaging will be done on day 2 or 3 of the menstrual cycle, trigger-shot and egg retrieval. — Functional Magnetic resonance imaging will be done on day 2 or 3 of the menstrual cycle, trigger-shot and egg retrieval.

SUMMARY:
The investigators aim is to investigate the brain's dynamic complexity across three phases of an ovarian stimulation cycle (basal, pre-OPU, mid-luteal), to observe the impact of externally administered hormones, and compare it with the corresponding phases of a natural menstrual cycle (early follicular, pre-ovulatory, mid-luteal) in the same woman. Brain activity patterns will be examined using resting-state fMRI in a sample of young, healthy, naturally cycling women.

DETAILED DESCRIPTION:
The investigators seeks to fill a significant gap in our understanding of the impact of ovarian stimulation on brain dynamics, an area that has not been previously explored. By investigating the brain's dynamic complexity across controlled ovarian stimulation cycle the investigators aim to shed light on how externally administered hormones influence brain activity patterns. Utilizing resting-state Functional Magnetic Resonance Imaging to examine a sample of young, healthy, naturally cycling women, this research will provide crucial insights into the safety and neurophysiological effects of ovarian stimulation. Understanding these effects is essential for ensuring the well-being of women undergoing oocyte freezing and other fertility treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 25 - 35 years old
* BMI: 20 - 30
* Anti-Mullerian Hormone (AMH): 1.3 - 5.9 ng/ml
* Regular Menstrual Cycle: 26-35 days
* In case of previous use of hormonal contraception: wash-out period of 3 month
* Meet standard safety and eligibility criteria for MRI scanning, including the absence of contraindications such as metallic implants, claustrophobia, or other medical conditions that preclude MRI

Exclusion Criteria:

* History of ovarian surgery
* Pathology of the ovaries
* Mental health disorders
* Use of medication influencing brain function
* Ongoing use of hormonal contraception (this would include OCP, but also patches and Mirena containing IUD)

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only naturally cycling women.
Study Population: Young (age range 25-35), healthy, naturally cycling women with a normal BMI, who want to undergo ovarian stimulation for oocyte vitrification.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Brain activity using functional magnetic resonance imaging (fMRI). | Measure at three cycle points: basal (day 2-3), ovulation (during ovulation or day after trigger-shot), and at luteal phase (7-10 days after ovulation or trigger shot).
  Comparison of brain activity between the natural menstrual cycle and a stimulated cycles using functional magnetic resonance imaging (fMRI) at three cycle points.

SECONDARY OUTCOMES:
Hormonal levels (Estradiol, LH, FSH, Progesterone) fluctuation. | Measure at three cycle points: basal (day 2-3), ovulation (during ovulation or day after trigger-shot), and at luteal phase (7-10 days after ovulation or trigger shot).
  Analyze relation of hormonal fluctuations (Estradiol, LH, FSH, Progesterone) at three cycle points with brain dynamics and neural connectivity.
Whole genome sequencing of patient. | Day 1 - baseline saliva sample collection.
  Sequence patient's genome using saliva sampling to observes the genetic basis of fertility traits, to identify genetic variants associated with various neural and fertility phenotypes.

CONTACTS AND LOCATIONS:
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

REFERENCES:
- [Background] Mueller JM, Pritschet L, Santander T, Taylor CM, Grafton ST, Jacobs EG, Carlson JM. Dynamic community detection reveals transient reorganization of functional brain networks across a female menstrual cycle. Netw Neurosci. 2021 Feb 1;5(1):125-144. doi: 10.1162/netn_a_00169. eCollection 2021. PMID 33688609
- [Background] Pritschet L, Santander T, Taylor CM, Layher E, Yu S, Miller MB, Grafton ST, Jacobs EG. Functional reorganization of brain networks across the human menstrual cycle. Neuroimage. 2020 Oct 15;220:117091. doi: 10.1016/j.neuroimage.2020.117091. Epub 2020 Jul 2. PMID 32621974